CLINICAL TRIAL: NCT02369354
Title: Transplant Social Worker Support for Live Kidney Donation in African Americans
Acronym: TALKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00052724; 1R01DK098759 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Results first posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Kidney Disease
Keywords: Kidney Transplant; African Americans
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Usual medical care at the Duke Kidney Transplant Clinic
- TALKS (Other): Usual Care plus TALKS Social Worker Intervention: Includes video, book, and Social Worker meetings
  Interventions: Behavioral: TALKS Social Worker Intervention
- TALKS PLUS (Other): Usual Care plus TALKS Social Worker Intervention: Includes video, book, and Social Worker meetings plus live donor financial assistance intervention
  Interventions: Behavioral: TALKS Social Worker Intervention; Other: Financial Assistance Intervention

INTERVENTIONS:
Behavioral: TALKS Social Worker Intervention — TALKS includes a video and book that describe patient and family experiences with talking about and considering live kidney transplantation. TALKS also includes a social worker meeting. Potential recipients meet with a transplant social worker for up to 60 minutes to identify potential barriers to considering or pursuing live donor kidney transplantation. They also are invited to have a second meeting with family and/or friends with the social worker for up to 60 minutes.
  Arms: TALKS; TALKS PLUS
Other: Financial Assistance Intervention — The financial assistance intervention offers potential donors the ability to draw from a "bank" of $2100 to reimburse their costs related to being evaluated for live kidney donation or for donating a kidney. Costs include, but are not limited to: child care, travel, time off work, and other out of pocket expenses related to being evaluated to become a live kidney donor or to donating.
  Arms: TALKS PLUS

SUMMARY:
Talking About Live Kidney Donation Support (TALKS) will study the effectiveness of education, behavior, and financial support interventions to improve consideration of live kidney transplantation/live kidney donation among African Americans on the deceased kidney waiting list. We hypothesize that interventions to help potential kidney transplant recipients and their potential donors overcome barriers to live donor kidney transplant (including family discussions, financial, or logistical barriers) could improve potential recipients' receipt of live kidney transplants. The main outcomes of TALKS will include whether potential recipients (1) have potential live donors call into the transplant center on their behalf; (2) have potential donors evaluated for transplant; or (3) receive a live donor kidney transplant.

DETAILED DESCRIPTION:
Live donor kidney transplantation (LDKT) represents an optimal therapy for many patients. However, African Americans have been persistently and significantly less likely to receive LDKT when compared to Whites. The process of seeking and establishing a live donor for LDKT requires potential donors overcome several potential obstacles to LKDT. As a critical first step to seeking LDKT, patients must engage their physicians and their family members or friends (who provide support for patients' health decisions and could also be potential donors) in discussions about LDKT to determine whether LDKT is a viable and/or desirable treatment option. LDKT discussions with physicians help patients and family members understand the risks and benefits of LDKT to both the potential recipient and any potential donors. Families' LDKT discussions help them establish whether it is possible to identify willing and medically eligible live donors, and they help families discuss the potential psychological, physical, and financial strains of LDKT on patients and families. Once discussions have occurred, potential donors must confront logistical (e.g., childcare or travel to transplant centers) and financial (e.g., unpaid time away from work) challenges associated with LDKT. Studies have shown that even when African American patients desire LDKT, rates of LDKT discussions are suboptimal. Further, African American potential live kidney donors are less likely than their White counterparts to complete the donor evaluation process, and they may be more sensitive than Whites to logistical and financial barriers to LDKT. Innovative strategies to overcome interpersonal, logistical and financial barriers to LDKT are sorely needed for African Americans, particularly those who may be highly motivated to seek this therapy. Transplant social workers routinely perform psychosocial evaluations on potential LDKT recipients and donors and are well suited to support families' navigation of LDKT discussions. Transplant social workers are also well versed in the financial aspects of LDKT (e.g., insurance coverage rules) and frequently provide financial guidance to potential LDKT recipients and donors. We will study innovative transplant social worker led interventions designed to help African American potential LDKT recipients and their families overcome interpersonal, logistical and financial barriers to LDKT. African Americans on the deceased kidney donor waiting list will be randomly assigned to (1) receive their usual care on the transplant list or (2) to one of two social worker led interventions-one which helps patients and families discuss LDKT with each other and with patients' physicians, and one which provides families with financial support to overcome logistical and financial barriers to LDKT. As a primary outcome, we will measure whether the interventions activate live kidney donation on African American potential recipients' behalf.

ELIGIBILITY:
For potential kidney transplant recipients (all arms):

Inclusion Criteria:

* Adult (18 yrs or older)
* African American
* Duke Kidney and Pancreas Transplant patients with end stage kidney disease
* Currently on the deceased donor kidney waiting list from the Duke Kidney and Pancreas Transplant Program
* Give consent to participate

Exclusion Criteria:

* Previous kidney transplant (Revised Sept 2016: persons who have previously received a deceased donor kidney transplant, but who have not previously received a live donor kidney transplant)
* Cognitively impaired/Change in cognition
* Impaired hearing or speech
* Non-English speaking

For family members or friends of potential kidney transplant recipients (TALK and TALK PLUS arms):

Inclusion Criteria:

* 18 or older
* Come to SWI meeting with patient
* Give consent to participate

For potential live kidney donors (TALKS PLUS arm only)

Inclusion Criteria:

* 18 or older
* Contact the study
* Give consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh E Boulware, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke School of Medicine, Division of General Internal Medicine, Durham, North Carolina, United States

REFERENCES:
- [Derived] Boulware LE, Sudan DL, Strigo TS, Ephraim PL, Davenport CA, Pendergast JF, Pounds I, Riley JA, Falkovic M, Alkon A, Hill-Briggs F, Cabacungan AN, Barrett TM, Mohottige D, McElroy L, Diamantidis CJ, Ellis MJ. Transplant social worker and donor financial assistance to increase living donor kidney transplants among African Americans: The TALKS Study, a randomized comparative effectiveness trial. Am J Transplant. 2021 Jun;21(6):2175-2187. doi: 10.1111/ajt.16403. Epub 2021 Jan 4. PMID 33210831
- [Derived] Strigo TS, Ephraim PL, Pounds I, Hill-Briggs F, Darrell L, Ellis M, Sudan D, Rabb H, Segev D, Wang NY, Kaiser M, Falkovic M, Lebov JF, Boulware LE. The TALKS study to improve communication, logistical, and financial barriers to live donor kidney transplantation in African Americans: protocol of a randomized clinical trial. BMC Nephrol. 2015 Oct 9;16:160. doi: 10.1186/s12882-015-0153-y. PMID 26452366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between September 2015 and May 2017. Participants were recruited from the Duke University Kidney and Pancreas Transplant Center in Durham, North Carolina. Transplant Center electronic health records were used to identify eligible patients.
Pre-assignment Details: Family members or friends of potential kidney transplant recipients and potential live kidney donors were not enrolled in the study.
Period: Overall Study
Arm/Group | Usual Care | TALKS | TALKS PLUS
Started | 100 | 100 | 100
Completed | 88 | 86 | 86
Not Completed | 12 | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | TALKS | TALKS PLUS | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 89 | 83 | 87 | 259
  >=65 years | 11 | 17 | 13 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.7 [43.3 to 59.6] | 52.3 [46.0 to 61.5] | 52.4 [45.5 to 60.9] | 52.3 [44.6 to 60.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 46 | 46 | 133
  Male | 59 | 54 | 54 | 167
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 100 | 100 | 100 | 300
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 100 | 100 | 300
Education [Count of Participants; unit: Participants]
  Intermediate or middle school (6-8) | 1 | 2 | 1 | 4
  High school (9-12) or GED | 37 | 38 | 38 | 113
  Two years of college | 30 | 30 | 33 | 93
  College | 22 | 25 | 18 | 65
  Graduate or professional school | 10 | 5 | 10 | 25
Employment [Count of Participants; unit: Participants]
  Full-time employee | 18 | 19 | 22 | 59
  Part-time employee | 6 | 10 | 5 | 21
  Student | 3 | 1 | 1 | 5
  Retired | 9 | 14 | 10 | 33
  Homemaker | 1 | 3 | 4 | 8
  Retired due to disability | 56 | 47 | 48 | 151
  Unemployed/looking for work | 6 | 6 | 10 | 22
  Refused | 1 | 0 | 0 | 1
Income [Count of Participants; unit: Participants]
  Under $20,000 | 18 | 18 | 22 | 58
  $20,000 - $39,999 | 21 | 24 | 25 | 70
  $40,000 - $59,999 | 26 | 14 | 20 | 60
  $60,000 or more | 22 | 26 | 19 | 67
  Refused/Don't know | 13 | 18 | 14 | 45
Poverty [Count of Participants; unit: Participants]
  Not in poverty | 70 | 65 | 67 | 202
  Near poverty | 7 | 9 | 8 | 24
  Poverty | 10 | 8 | 11 | 29
  Missing | 13 | 18 | 14 | 45
Medical Insurance [Count of Participants; unit: Participants]
  Private | 22 | 23 | 23 | 68
  Medicaid Only | 5 | 2 | 6 | 13
  Medicare Only | 57 | 53 | 48 | 158
  Medicare/Medicaid | 14 | 21 | 22 | 57
  Other | 2 | 1 | 1 | 4
Marital status [Count of Participants; unit: Participants]
  Married/living with partner | 48 | 44 | 44 | 136
  Separated | 3 | 7 | 8 | 18
  Divorced | 18 | 8 | 14 | 40
  Single, never married | 27 | 29 | 33 | 89
  Widowed | 4 | 12 | 1 | 17
Family members [Count of Participants; unit: Participants]
  Has child(ren): Yes | 77 | 85 | 78 | 240
  Has child(ren): No | 23 | 15 | 22 | 60
  Has sibling(s): Yes | 86 | 91 | 91 | 268
  Has sibling(s): No | 14 | 9 | 9 | 32
  Mother living: Yes | 43 | 50 | 55 | 148
  Mother living: No | 57 | 50 | 45 | 152
  Father living: Yes | 35 | 23 | 31 | 89
  Father living: No | 65 | 77 | 69 | 211
Total potential immediate family donors [Median (Inter-Quartile Range); unit: potential immediate family donors] | 6 [4 to 8] | 6 [4 to 8] | 5.5 [4 to 8] | 6 [4 to 8]
Family history of kidney disease [Count of Participants; unit: Participants] | 52 | 49 | 51 | 152
Health literacy [Count of Participants; unit: Participants]
  ≤3rd grade | 3 | 3 | 4 | 10
  4th-6th grade | 5 | 4 | 4 | 13
  7th-8th grade | 27 | 29 | 33 | 89
  ≥9th grade | 64 | 58 | 55 | 177
  Missing | 1 | 6 | 4 | 11
Years on the waiting list [Median (Inter-Quartile Range); unit: years] | 0.5 [0.2 to 1.8] | 0.8 [0.2 to 1.9] | 0.9 [0.2 to 2.1] | 0.8 [0.2 to 1.9]
Current end-stage (ESRD) renal disease treatment [Count of Participants; unit: Participants]
  No kidney replacement treatment yet | 15 | 16 | 22 | 53
  In-center hemodialysis | 63 | 63 | 63 | 189
  Home hemodialysis | 6 | 3 | 3 | 12
  Peritoneal dialysis | 16 | 18 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Live Kidney Donor Activation Events
Description: Composite rate of live kidney donor inquiries on behalf of participants, completed live kidney donor transplant evaluations, and live kidney donor transplants in each arm, ascertained via medical records maintained by the Duke Kidney and Pancreas Transplant Program.
Time Frame: 24 months post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | TALKS | TALKS PLUS
Number analyzed (Participants) | 100 | 100 | 100
Participants
  0 Activation events | 87 | 86 | 88
  1 Activation event | 5 | 4 | 7
  2 Activation events | 3 | 7 | 2
  3 Activation events | 3 | 2 | 3
  4 Activation events | 1 | 1 | 0
  >=5 Activation events | 1 | 0 | 0

2. Secondary Outcome: Number of Participants With Potential Recipient Interest and Pursuit of Live Donor Kidney Transplantation
Description: Potential kidney recipients' behaviors reflecting their interest and pursuit of live donor kidney transplantation, including: self-reported live donor kidney transplant discussions with physicians, self-reported live donor kidney transplant discussions with family, and identification of a potential live donor.
Time Frame: 24 months post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | TALKS | TALKS PLUS
Number analyzed (Participants) | 100 | 100 | 100
Participants
  Low pursuit (did not discuss with family) | 1 | 0 | 1
  Moderate (Discussed with family) | 12 | 10 | 8
  High (Identified potential donor) | 58 | 57 | 64
  Data missing | 29 | 33 | 27

3. Secondary Outcome: Number of Participants With Live Donor Evaluations
Description: Passive follow up of participants for 2 years to assess completed live kidney donor transplant evaluations in each arm, ascertained via medical records maintained by the Duke Kidney and Pancreas Transplant Program.
Time Frame: 24 months post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | TALKS | TALKS PLUS
Number analyzed (Participants) | 100 | 100 | 100
Participants
  0 Evaluations | 93 | 93 | 97
  1 Evaluation | 5 | 7 | 3
  2 Evaluations | 2 | 0 | 0
  3 Evaluations | 0 | 0 | 0
  4 Evaluations | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Live Kidney Donor Transplants
Description: Passive follow up of participants for 2 years to assess live kidney donor transplants in each arm, ascertained via medical records maintained by the Duke Kidney and Pancreas Transplant Program.
Time Frame: 24 months post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | TALKS | TALKS PLUS
Number analyzed (Participants) | 100 | 100 | 100
Participants | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: 24 months post randomization
Arm/Group | Usual Care | TALKS | TALKS PLUS
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100

LIMITATIONS AND CAVEATS:
The study was performed at a single transplant center, which may limit generalizability of results. The study's follow-up time may not have been sufficient for participants to identify new potential donors, initiate discussions, and for potential donors to become activated toward living kidney donation. Additionally, participants with longer wait-list times may have been less motivated to pursue LDKT. Lastly, we did not assess reasons for non-use of the TALKS financial assistance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02369354/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02369354/SAP_001.pdf